CLINICAL TRIAL: NCT03281954
Title: A Randomized, Double-Blind, Phase III Clinical Trial of Neoadjuvant Chemotherapy With Atezolizumab or Placebo in Patients With Triple-Negative Breast Cancer Followed by Adjuvant Continuation of Atezolizumab or Placebo
Brief Title: Clinical Trial of Neoadjuvant Chemotherapy With Atezolizumab or Placebo in Patients With Triple-Negative Breast Cancer Followed After Surgery by Atezolizumab or Placebo
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: Genentech, Inc. (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NSABP B-59/GBG 96-GeparDouze; 2017-002771-25 (EudraCT Number); MO39875 (Other: Genentech, Inc.)
Record Dates: First submitted 2017-09-08; First posted 2017-09-13 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Triple Negative Breast Cancer
Keywords: anti-PD-L1 antibody; TNBC
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — atezolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): IV infusion once every 3 weeks for 4 doses (Cycle 1), once every 3 weeks for 4 doses (Cycle 2) and once every 3 weeks after surgery for 1 year after first dose
  Interventions: Drug: Placebo
- Atezolizumab (Experimental): IV infusion, 1200mg, once every 3 weeks for 4 doses (Cycle 1), once every 3 weeks for 4 doses (Cycle 2) and once every 3 weeks after surgery for 1 year after first dose
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Placebo — Following randomization, patients will receive Paclitaxel 80 mg/m2 IV weekly x 12 doses + Carboplatin AUC of 5 IV Day 1 every 3 weeks for 4 cycles + placebo IV Day 1 every 3 weeks for 4 doses.
  Followed 2-3 weeks later by Doxorubicin (A) 60 mg/m2 IV + cyclophosphamide (C) 600 mg/m2 IV Day 1 every 2 or 3 weeks for 4 cycles OR Epirubicin (E) 90 mg/m2 IV + cyclophosphamide (C) 600 mg/m2 IV Day 1 every 2 or 3 weeks for 4 cycles.
  + placebo IV Day 1 every 3 weeks for 3 to 4 doses depending on AC/EC schedule used.
  Approximately 3-4 weeks later: Surgery (Lumpectomy or mastectomy and axillary staging), followed by placebo IV Day 1 every 3 weeks after surgery until 1 year after the first dose.
  Arms: Placebo
Drug: Atezolizumab — Following randomization, patients will receive Paclitaxel 80 mg/m2 IV weekly x 12 doses + Carboplatin AUC of 5 IV Day 1 every 3 weeks for 4 cycles + Atezolizumab 1200 mg Day 1 every 3 weeks for 4 doses.
  Followed 2-3 weeks later by Doxorubicin (A) 60 mg/m2 IV + cyclophosphamide (C) 600 mg/m2 IV Day 1 every 2 or 3 weeks for 4 cycles OR Epirubicin (E) 90 mg/m2 IV + cyclophosphamide (C) 600 mg/m2 IV Day 1 every 2 or 3 weeks for 4 cycles.
  + Atezolizumab 1200 mg Day 1 every 3 weeks for 3 to 4 doses depending on AC/EC schedule used.
  Approximately 3-4 weeks later: Surgery (Lumpectomy or mastectomy and axillary staging), followed by Atezolizumab 1200 mg Day 1 every 3 weeks after surgery until 1 year after the first dose.
  Arms: Atezolizumab

SUMMARY:
The main purpose of this study is to learn if the usual chemotherapy given before surgery (neoadjuvant therapy) for breast cancer plus the experimental drug, atezolizumab, is better than the usual chemotherapy plus a placebo. (A placebo is a drug that looks like the study drug but contains no medication.) The usual chemotherapy in this study is paclitaxel (WP) and carboplatin followed by doxorubicin and cyclophosphamide (AC) or epirubicin and cyclophosphamide (EC). Usually, after neoadjuvant therapy and surgery for triple negative breast cancer, no additional treatment is given unless the cancer returns. This study will also look at continuing treatment after surgery with atezolizumab or the placebo. To be better, atezolizumab given with the neoadjuvant therapy should be better at: 1) decreasing the amount of tumor in the breast than the placebo given with the usual chemotherapy and 2) decreasing the chance of the cancer from returning after surgery.

Another purpose of this study is to test the good and bad effects of atezolizumab when added to the usual chemotherapy. Atezolizumab may keep your cancer from growing but it can also cause side effects.

DETAILED DESCRIPTION:
NSABP B-59/GBG 96-GeparDouze is a prospective, randomized, double-blind, Phase III clinical trial. This is a collaborative study being conducted by NSABP Foundation, Inc. in partnership with the German Breast Group (GBG), and supported by funding by Genentech, a Member of the Roche Group, and F. Hoffmann-La Roche, Ltd.

In this clinical trial of neoadjuvant and adjuvant administration of atezolizumab/placebo in patients with high risk triple-negative breast cancer, the potential incremental efficacy and safety of neoadjuvant administration of atezolizumab/placebo with a sequential regimen of weekly paclitaxel with every-3-week carboplatin followed immediately by neoadjuvant administration of atezolizumab/placebo with AC/EC will be evaluated. Patients will then undergo surgery. Following recovery from surgery, patients will initiate approximately 6 months of adjuvant therapy with atezolizumab/placebo and receive the same investigational agent they received pre-operatively. Administration of radiation therapy will be based on local standards at the discretion of patients and investigators, but if administered, atezolizumab/placebo will be administered concurrently. Adjuvant atezolizumab/placebo may be delayed until after completion of radiation therapy per investigator discretion. Patients with residual invasive cancer at the time of surgery may receive capecitabine concurrently with atezolizumab/placebo in the adjuvant setting per investigator discretion and local guidelines. Patients with germline BRCA1 or BRCA2 mutations with residual invasive cancer at the time of surgery may receive olaparib in the adjuvant setting per investigator discretion and local guidelines. Patients receiving olaparib must discontinue atezolizumab/placebo.

The primary aims of the study are 1) to determine value of atezolizumab in improving pathologic complete response in the breast and post-therapy lymph nodes evaluated histologically (pCR breast and nodes [(ypT0/Tis ypN0)]), and 2) to determine the value of atezolizumab in improving event-free survival (EFS). Secondary aims include: pathologic complete response in the breast (ypT0/Tis); pathologic complete response in the breast and lymph nodes (ypT0 ypN0); positive nodal status conversion rate; overall survival; recurrence-free interval: distant disease-free survival; brain metastases free survival; and toxicity. The stratification factors for the study are: 1) clinical size of the primary tumor (1.1-3.0 cm; > 3.0 cm); 2) nodal status as determined by protocol-specified criteria (negative, positive); 3) AC/EC (every 2 weeks; every 3 weeks); and 4) Region (North America; Europe).

For patient eligibility, local testing on the diagnostic core must have determined the patient's tumor to be ER-negative, PgR-negative, and HER2-negative by current ASCO/CAP guidelines. Material from either the diagnostic core biopsy or the research biopsy must be sent for central testing for confirmation of ER, PgR, and HER2 to confirm eligibility. If local testing has determined a tumor to be HER2 equivocal or to have a borderline ER/PgR status (% IHC staining < 10% for both), material may be submitted for central testing to determine eligibility.

In order to proactively identify and further assess any cardiac toxicity that may occur with the combination of anthracyclines and atezolizumab, this study includes a cardiac safety lead-in for the first 60 patients who initiate AC/EC. The safety lead-in will consist of assessment of ECG and serum troponin-T obtained just prior to administration of the first dose of AC/EC, following completion of the administration of the 1st and 3rd cycle of AC/EC prior to initiation of the atezolizumab/placebo. An additional assessment of LVEF with echocardiogram or MUGA scan will also be obtained prior to the 3rd dose of AC/EC. In order to provide an early assessment of cardiac safety, results of the troponin-T assessments, ECGs, LVEF assessment, and cardiac safety data will be evaluated by the Data Safety Monitoring Board (DSMB) when the last of the initial 20 patients who initiate AC/EC undergo their scheduled post-surgery LVEF assessment. When the last of the first 60 patients to initiate AC/EC undergo their scheduled post-surgery LVEF assessment, results of the troponin assessments, ECGs, LVEF assessments, and cardiac safety data from all 60 patients will be evaluated by the DSMB.

Research core biopsies of breast primary at baseline and 1-4 days prior to the second dose of atezolizumab/placebo are a study requirement for all patients. One to three representative blocks of residual primary tumor containing the maximum amount of tumor and node with the largest focus of metastasis is required from the definitive breast surgery if gross residual disease is greater than or equal to 1.0 cm. If gross residual disease is less than 1.0 cm, tissue should be submitted, if possible. Blood specimens will be collected on all patients at baseline for exploratory biomarker analysis and to support future correlative studies.

Accrual to NSABP B-59/GBG 96-GeparDouze began in December 2017 and was completed in May 2021 with a total of 1550 patients randomized. Based on actual accrual and the decision to eliminate pCR as a co-primary endpoint, we recalculated the power to detect a hazard ratio of 0.70 attributed to the addition of atezolizumab, assuming a lost-to-follow-up rate of 0.00083 per month, using the actual accrual pattern for the power calculation. With 1550 patients accrued in 42 months, an additional 22 months follow up will allow us to obtain 252 events under the assumptions stated above, which will provide 80% power to detect a HR of 0.7 between the atezolizumab and the placebo arm at an overall 2-sided alpha level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have consented to participate and, prior to beginning specific study procedures, must have signed and dated an appropriate IRB-approved consent form that conforms to federal and institutional guidelines for study treatment and for submission of tumor samples from a research biospy as required by NSABP B-59/GBG 96-GeparDouze for baseline correlative science studies.
* The diagnosis of invasive adenocarcinoma of the breast must have been made by core needle biopsy.
* Local testing on the diagnostic core must have determined the tumor to be ER-negative, PgR-negative, and HER2-negative by current ASCO/CAP guidelines. (If local testing has determined a tumor to be HER2 equivocal or to have a borderline ER/PgR status (% IHC staining < 10% for both) and other eligibility criteria are met, material may be submitted for central testing to determine eligibility.)
* Central testing for ER, PgR, and HER2 will be performed, and the tumor must be determined to be ER-negative, PgR-negative, and HER2-negative by current ASCO/CAP Guidelines Recommendations.
* The tumor specimen used for central ER, PgR, and HER2 testing must also be used for central testing of PD-L1 status using the Ventana PD-L1 testing result including PD-L1 indeterminate Patients will be classifies as positive, negative, or indeterminate for stratification purposes.
* Patients must be ≥ 18 years old.
* Patient may be female or male.
* The ECOG performance status must be 0-1.
* The primary tumor can be clinical stage T2 or T3, if clinically node negative according to AJCC 7th Edition. If the regional lymph nodes are cN1 and cytologically or histologically positive or cN2-N3 with or without a biopsy, the primary breast tumor can be clinically T1c, T2, or T3.
* Ipsilateral axillary lymph nodes must be evaluated by imaging (mammogram, ultrasound, and/or MRI) within 84 days prior to study entry. If suspicious or abnormal, FNA or core biopsy is recommended. Findings of these evaluations will be used to define the nodal status prior to study entry according to the following criteria:

  * Nodal status - negative (Imaging of the axilla is negative; Imaging is suspicious or abnormal but the FNA or core biopsy of the questionable node[s] on imaging is negative)
  * Nodal status - positive (FNA or core biopsy of the node[s] is cytologically or histologically suspicious or positive; Imaging is suspicious or abnormal but FNA or core biopsy was not performed.)
* Patients with synchronous bilateral or multicentric HER2-negative breast cancer are eligible as long as the highest risk tumor is ER-negative and PgR-negative and meets stage eligibility criteria. All of the other invasive tumors must also be HER2-negative by ASCO/CAP Guidelines based on local testing. Central testing to confirm TNBC status is only required for the highest risk tumor.
* Blood counts performed within 28 days prior to randomization must meet the following criteria:

  * ANC must be ≥ 1500/mm3;
  * platelet count must be ≥ 100,000/mm3; and
  * hemoglobin must be ≥10 g/dL.
* The following criteria for evidence of adequate hepatic function performed within 28 days prior to randomization must be met:

  * total bilirubin must be ≤ ULN for the lab unless the patient has a bilirubin elevation > ULN to 1.5 x ULN due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin; and
  * alkaline phosphatase must be ≤ 2.5 x ULN for the lab; and
  * AST and ALT must be ≤ 1.5 x ULN for the lab.
* Patients with AST or ALT or alkaline phosphatase > ULN are eligible for inclusion in the study if liver imaging (CT, MRI, abdominal ultrasound, PET-CT, or PET scan) performed within 28 days prior to randomization does not demonstrate metastatic disease and the requirements in criterion (just above) are met.
* Patients with alkaline phosphatase that is > ULN but less than or equal to 2.5 x ULN or with unexplained bone pain are eligible for inclusion in the study if bone imaging (bone scan, PET-CT scan, or PET scan) supported by additional studies when indicated (CT, x-ray, MRI) performed within 28 days prior to randomization does not demonstrate metastatic disease.
* Patients with N2 or N3 nodal disease or T3 primary disease must undergo liver and bone imaging (as described in 4.1.13 and 4.1.14) within 28 days prior to randomization, irrespective of baseline lab results, and studies must not demonstrate metastatic disease. Chest imaging with chest x-ray PA and Lateral, CT of the chest, or PET-CT must also be performed.
* Creatinine clearance ≥ 50 mL/min (see Section 7.2.1 for instructions regarding calculation of creatinine clearance) performed within 28 days prior to randomization.
* PT/INR ≤ ULN within 28 days of randomization. Patients receiving therapeutic anti-coagulants are not eligible.
* A serum TSH and AM (morning) cortisol performed within 28 days prior to randomization to obtain a baseline value. Patients with abnormal TSH or AM cortisol baseline levels should be further evaluated and managed per institutional standards. Asymptomatic patients who require initiation or adjustment of medication or are followed without initiating treatment based on endocrinologist's recommendations are eligible.
* LVEF assessment must be performed within 42 days prior to randomization. (LVEF assessment performed by echocardiogram is preferred; however, MUGA scan may be substituted based on institutional preferences.) The LVEF must be ≥ 55% regardless of the cardiac imaging facility's lower limit of normal.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 5 months after the last dose of atezolizumab/placebo or 12 months after the last dose of chemotherapy.

  * A woman is considered to be of childbearing potential if she is not postmenopausal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).
  * Examples of contraceptive methods with a failure rate of < 1% per year include: bilateral tubal ligation; male partner sterilization; hormonal contraceptives that inhibit ovulation; hormone-releasing intrauterine devices; copper intrauterine devices.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
* Patient must be willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Excisional biopsy or lumpectomy performed prior to study entry.
* FNA alone to diagnose the breast cancer.
* Surgical axillary staging procedure prior to randomization. Exception: FNA or core biopsy of an axillary node is permitted for any patient. A pre-neoadjuvant therapy sentinel lymph node biopsy for patients with clinically negative axillary nodes is prohibited.
* Definitive clinical or radiologic evidence of metastatic disease.
* Previous history of contralateral invasive breast cancer. (Patients with synchronous and/or previous contralateral DCIS or LCIS are eligible.)
* Previous history of ipsilateral invasive breast cancer or ipsilateral DCIS. (Patients with synchronous or previous ipsilateral LCIS are eligible.)
* History of non-breast malignancies (except for in situ cancers treated only by local excision and basal cell and squamous cell carcinomas of the skin) within 5 years prior to study entry.
* Treatment including radiation therapy, chemotherapy, or targeted therapy, for the currently diagnosed breast cancer prior to randomization.
* Previous therapy with anthracyclines or taxanes for any malignancy.
* Cardiac disease (history of and/or active disease) that would preclude the use of the drugs included in the treatment regimens. This includes but is not confined to:

  * Active cardiac disease: angina pectoris that requires the use of anti-anginal medication; ventricular arrhythmias except for benign premature ventricular contractions; supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication; conduction abnormality requiring a pacemaker; valvular disease with documented compromise in cardiac function; or symptomatic pericarditis.
  * History of cardiac disease: myocardial infarction documented by elevated cardiac enzymes or persistent regional wall abnormalities on assessment of left ventricular function within 6 months prior to randomization; history of documented CHF; or documented cardiomyopathy.
* Uncontrolled hypertension defined as sustained systolic BP > 150 mmHg or diastolic BP > 90 mmHg. (Patients with initial BP elevations are eligible if initiation or adjustment of BP medication lowers pressure to meet entry criteria.) Patients requiring ≥ 3 BP medications are not eligible.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
* Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells.
* Known allergy or hypersensitivity to the components of the atezolizumab formulation.
* Known allergy or hypersensitivity to the components of the doxorubicin, epirubicin, cyclophosphamide, carboplatin, or paclitaxel formulations.
* Known allergy or hypersensitivity to liposomal or pegylated G-CSF formulations.
* Active or history of autoimmune disease or immune deficiency, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis for a more comprehensive list of autoimmune diseases and immune deficiencies) with the following exceptions:

  * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for this study.
  * Patients with controlled Type 1 diabetes mellitus on a stable dose of insulin regimen may be eligible for this study.
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are permitted provided all of following conditions are met: Rash must cover < 10% of body surface area; Disease is well controlled at baseline and requires only low-potency topical corticosteroids; No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
* Patients known to be HIV positive.
* Active hepatitis B virus (HBV) infection, defined as having a positive hepatitis B surface antigen (HBsAg) test at screening. Patients with a past or resolved HBV infection, defined as having a negative HBsAg test and a positive total hepatitis B core antibody (HBcAb) test at screening, are eligible for the study if active HBV infection is ruled out on the basis of HBV DNA viral load per local guidelines.
* Active hepatitis C virus (HCV) infection, defined as having a positive HCV antibody test at screening confirmed by a polymerase chain reaction (PCR) positive for HCV RNA.
* Patients with clinically active tuberculosis.
* Severe infection within 28 days prior to randomization, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
* Prior allogeneic stem cell or solid organ transplantation.
* Administration of a live, attenuated vaccine within 28 days prior to randomization or anticipation that such vaccine will be required during the study. Patients must agree not to receive live, attenuated influenza vaccine (e.g., FluMist) within 28 days prior to randomization, during treatment or within 5 months following the last dose of atezolizumab/placebo.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.
* Prior treatment with CD137 agonists or immune checkpoint-blockade therapies, including anti-CD40, anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies.
* Treatment with systemic immunosuppressive medications (including but not limited to interferons, IL-2) within 28 days or 5 half-lives of the drug, whichever is longer, prior to randomization.
* Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis [anti-TNF] factor agents) within 14 days prior to randomization or anticipation of need for systemic immunosuppressive medications during the study.
* Nervous system disorder (paresthesias, peripheral motor neuropathy, or peripheral sensory neuropathy) ≥ Grade 2, per the CTCAE v4.0.
* Symptomatic peripheral ischemia.
* Pregnancy or lactation at the time of randomization or intention to become pregnant during the study. (Note: Negative serum pregnancy test must be obtained within 14 days prior to randomization).
* Use of any investigational agent within 28 days prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1550 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | From randomization until event, through study follow up to the time target number of events is obtained, up to 5 years
  Time from randomization until event

SECONDARY OUTCOMES:
Overall survival (OS) | From date of randomization through study follow-up, to the time the target number of events is obtained, up to 5 years
  Time from randomization until death from any cause
Pathologic complete response in the breast and lymph nodes (ypT0/Tis ypN0) | Following completion of neoadjuvant therapy (ypT0/Tis ypN0)
  Absence of any invasive component in the resected breast specimen and all resected lymph nodes
Distant disease-free survival (DDFS) | From date of randomization through study follow-up, to the time the target number of events is obtained, up to 5 years
  Time from randomization until distant recurrence, death from breast cancer, death from other causes, and second primary invasive cancer (non-breast)
Disease-free survival (DFS) | From the first breast surgical procedure to the first disease recurrence or death from any cause
  Ipsilateral invasive breast tumor recurrence, ipsilateral local-regional invasive breast cancer recurrence, distant recurrence, contralateral invasive breast cancer, ipsilateral or contralateral DCIS, second primary non-breast invasive cancer and death attributable to any cause including breast cancer, non-breast cancer, or unknown cause.
Frequency of Adverse Events | From beginning of study therapy to 90 days after last dose of study therapy
  Frequency of adverse events graded according to the NCI Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0)
Frequency of immune Adverse Events of Special Interest | From beginning of study therapy to 90 days after last dose of study therapy
  Frequency of immune adverse events of special interest according to the NCI Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0)
Cardiac safety lead-in (Troponin-T) | prior to initial dose of AC/EC following completion of carboplatin/paclitaxel co-administered with atezolizumab/placebo, approximately 12 weeks
  Troponin-T levels in blood prior to initial dose of AC/EC following completion of carboplatin/paclitaxel co-administered with atezolizumab/placebo
Cardiac safety lead-in (Troponin-T) | After administration of the 1st dose of AC/EC prior to administration of atezolizumab/placebo, approximately 1 hour after beginning the 1st dose of AC/EC
  Troponin-T levels in blood after administration of the 1st cycle of AC/EC prior to administration of atezolizumab/placebo
Cardiac safety lead-in (Troponin-T) | After administration of the 3rd dose (Cycle 3; each cycle is 21 days) of AC/EC prior to administration of atezolizumab/placebo, approximately 1 hour after beginning the 3rd dose of AC/EC
  Troponin-T levels in blood after administration of the 3rd cycle of AC/EC prior to administration of atezolizumab/placebo
Cardiac safety lead-in (Left ventricular ejection fraction; LVEF) | Prior to initiation of carboplatin/paclitaxel and atezolizumab/placebo, at baseline
  LVEF levels measured at baseline prior to initiation of carboplatin/paclitaxel and atezolizumab/placebo
Cardiac safety lead-in (Left ventricular ejection fraction; LVEF) | Prior to the 3rd cycle (each cycle is every 21 days) of AC/EC, approximately 6 weeks after initiation of AC/EC
  LVEF levels measured before 3rd cycle of AC/EC
Cardiac safety lead-in (Left ventricular ejection fraction; LVEF) | Four to 6 weeks after surgery
  LVEF levels measured after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSBP Foundation, Inc.
Locations (217):
- United States (212):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Katmai Oncology Group, Anchorage, Alaska
  - St. Bernard's Medical Center, Jonesboro, Arkansas
  - St. Bernard's Medical Center, Paragould, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Arrowhead Regional Medical Center, Colton, California
  - City of Hope, Duarte, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - Kaiser Permanente-Sunset, Los Angeles, California
  - Kaiser Permanente-West Los Angeles, Los Angeles, California
  - Kaiser Permanente-Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente Medical Group, San Diego, California
  - Kaiser Permanente-Zion, San Diego, California
  - Kaiser Permanente - Otay, San Diego, California
  - Kaiser Permanente- San Marcos, San Marcos, California
  - City of Hope - South Pasadena, South Pasadena, California
  - Torrance Memorial Physician Network, Torrance, California
  - City of Hope - Upland, Upland, California
  - PIH Health, Whittier, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Mount Sinai Comprehensive Cancer Center Aventura, Aventura, Florida
  - Memorial Healthcare System Office of Human Research, Hollywood, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - UF Health Cancer Center at Orlando Health, Orlando, Florida
  - Gwinnett Hospital System Center for Cancer Care, Duluth, Georgia
  - Gwinnett Hospital System Center for Cancer Care, Lawrenceville, Georgia
  - Gwinnett Hospital System Center for Cancer Care, Snellville, Georgia
  - Illinois Cancer Care-Bloomington, Bloomington, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Affiliated Oncologists, Chicago Ridge, Illinois
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Emhurst Memorial Nancy W. Knowles Cancer Center, Elmhurst, Illinois
  - Illinois Cancer Care-Galesburg, Galesburg, Illinois
  - Edward Cancer Center, Naperville, Illinois
  - Illinois Cancer Care-Ottawa, Ottawa, Illinois
  - Illinois Cancer Care PC, Peoria, Illinois
  - Illinois Cancer Care-Peru, Peru, Illinois
  - Edward Cancer Center Plainfield, Plainfield, Illinois
  - Cancer Care Specialists of Central Illinois-Swansea, Swansea, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc (W. Jefferson Blvd), Fort Wayne, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc (Parkview Plaza), Fort Wayne, Indiana
  - Mercy Medical Center Hall-Perrine Cancer Center, Cedar Rapids, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Susan B. Allen Memorial Hosptial, El Dorado, Kansas
  - Cancer Center at Mercy - W. Laurel, Independence, Kansas
  - Kingman Community Hospital, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - McPherson Center for Health, McPherson, Kansas
  - Newton Medical Center, Newton, Kansas
  - Labette Health, Parsons, Kansas
  - Pratt Regional Medical Center, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - Winfield Healthcare Center, Winfield, Kansas
  - Norton Cancer Institute-Downtown, Louisville, Kentucky
  - Norton Cancer Institute-Norton Healthcare Pavilion, Louisville, Kentucky
  - University of Louisville-James Graham Brown Cancer Center, Louisville, Kentucky
  - Baptist Health Louisville; Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Norton Cancer Institute-St Matthews, Louisville, Kentucky
  - Norton Cancer Institute-Brownsboro, Louisville, Kentucky
  - Ochsner Medical Center-Kenner, Kenner, Louisiana
  - West Jefferson Medical Center Cancer Center, Marrero, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Medstar Union Memorial Hospital, Baltimore, Maryland
  - Harry and Jeanette Weinberg Cancer Center at Franklin Square, Baltimore, Maryland
  - Maryland Oncology Hematology, Bethesda, Maryland
  - Maryland Oncology - Hematology Brandywine, Brandywine, Maryland
  - Maryland Oncology - Hematology PA, Columbia, Maryland
  - Maryland Oncology - Hematology Frederick, Frederick, Maryland
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - Maryland Oncology - Hematology PA, Lanham, Maryland
  - Maryland Oncology Hematology, Rockville, Maryland
  - Capital Hematology Oncology Associates, Silver Spring, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - University of Maryland, St. Joseph Medical Center, Towson, Maryland
  - Maryland Oncology Hematology, Wheaton, Maryland
  - Berkshire Hematology Oncology Services at Berkshire Medical Center Cancer and Infusion Center, Pittsfield, Massachusetts
  - Henry Ford Cancer Institute Brownstown, Brownstown, Michigan
  - Henry Ford Cancer Institute Macomb Hospital, Clinton Township, Michigan
  - Henry Ford Medical Center Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Henry Ford Allegiance Health, Jackson, Michigan
  - Michigan State University-Breslin Cancer Center, Lansing, Michigan
  - Henry Ford Medical Center Columbus, Novi, Michigan
  - Henry Ford Hospital W Bloomfield, West Bloomfield, Michigan
  - Henry Ford Cancer Institute Wyandotte Hospital, Wyandotte, Michigan
  - University of Missouri-Ellis Fischel Cancer Center, Columbia, Missouri
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - MD Anderson Cancer Center at Cooper, Voorhees Township, New Jersey
  - New York Oncology Hematology PC, Albany, New York
  - Broome Oncolgy, Binghamton, New York
  - Broome Oncology, Johnson City, New York
  - Health Quest Medical Practice, Poughkeepsie, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - RHOA of Cary, Cary, North Carolina
  - Waverly Hematology Oncology, Cary, North Carolina
  - Carolinas Medical Center-Levine Cancer Insitute, Charlotte, North Carolina
  - Levine Cancer Center Institute Pineville, Charlotte, North Carolina
  - RHOA of Garner, Garner, North Carolina
  - UNC Regional Physicians Hematology and Oncolgoy, High Point, North Carolina
  - FirstHealth of the Carolinas FirstHealth Outpatient Cancer Center, Pinehurst, North Carolina
  - Rex Cancer Center, Raleigh, North Carolina
  - RHOA of Blue Ridge, Raleigh, North Carolina
  - RCC of Wakefield, Raleigh, North Carolina
  - Nash UNC Health Care - Danny Talbott Cancer Center, Rocky Mount, North Carolina
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Aultman Alliance Cancer Center, Alliance, Ohio
  - Aultman Hospital, Canton, Ohio
  - Aultman Medical Group Hematology and Oncology, Canton, Ohio
  - The Ohio State University Wexner Medical Center-Investigational Drug Service Oncology, Columbus, Ohio
  - The Stephanie Speilman Comprehensive Breast Center, Columbus, Ohio
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Kaiser Permanente Northwest-Oncology/Hematology, Portland, Oregon
  - Northwest Cancer Specialists, Tigard, Oregon
  - UPMC Hillman Cancer Center-Beaver, Beaver, Pennsylvania
  - UPMC Hillman Cancer Center - Passavant North, Cranberry Township, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Allegheny Cancer Institute St. Vincent, Erie, Pennsylvania
  - St. Vincent Hospital, Erie, Pennsylvania
  - UPMC Cancer Center Horizon, Farrell, Pennsylvania
  - Wellspan Medical Oncology, Gettysburg, Pennsylvania
  - UPMC Hillman Cancer Center- Mountain View, Greensburg, Pennsylvania
  - UPMC Cancer Center Greenville, Greenville, Pennsylvania
  - AHN Cancer Institute at Jefferson, Jefferson Hills, Pennsylvania
  - Seechler Family Cancer Center, Lebanon, Pennsylvania
  - Forbes Regional Hospital, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center UPMC East-Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center Norwin, N. Huntingdon, Pennsylvania
  - UPMC Hillman Cancer Center New Castle, New Castle, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - WPAON at AGH, Pittsburgh, Pennsylvania
  - WPAON at WPH, Pittsburgh, Pennsylvania
  - Magee-Women's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - UPCI Investigational Drug Services, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center @ Passavant - HOA, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center @ Passavant - OHA, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center-Upper Saint Clair, Pittsburgh, Pennsylvania
  - UPMC Cancer Center Northwest, Seneca, Pennsylvania
  - UPMC Hillman Cancer Center - Uniontown, Uniontown, Pennsylvania
  - UPMC Hillman Cancer Center-Washington, Washington, Pennsylvania
  - Wexford Health & Wellness Pavilion, Wexford, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - Wellspan Health-York Cancer Center Oncology Research, York, Pennsylvania
  - Women's and Infants Hospital, Providence, Rhode Island
  - Gibbs Cancer Center and Research Institute - Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute-Sioux Falls, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Wellmont Cancer Institute, Johnson City, Tennessee
  - Wellmont Cancer Institute, Kingsport, Tennessee
  - Dell Seton Medical Center at the University of Texas-Seton Infusion Center, Austin, Texas
  - Texas Oncology Bedford, Bedford, Texas
  - Texas Oncology Carrollton, Carrollton, Texas
  - Texas Oncology - Methodist Dallas Cancer Center, Dallas, Texas
  - Texas Oncology - Medical City Dallas, Dallas, Texas
  - Texas Oncology Dallas Presbyterian Hospital, Dallas, Texas
  - Texas Oncology Denton, Denton, Texas
  - Texas Oncology Flower Mound, Flower Mound, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Cancer Center, Houston, Texas
  - Harris Health System-Smith Clinic, Houston, Texas
  - Texas Oncology - McAllen South Second, McAllen, Texas
  - Texas Oncology Midland Allison Cancer Center, Midland, Texas
  - Texas Oncology Plano, Plano, Texas
  - Texas Oncology - The Woodlands, The Woodlands, Texas
  - Wellmont Medical Associates-Oncology and Hematology, Bristol, Virginia
  - Virginia Cancer Care Specialist, Leesburg, Virginia
  - Centra Lynchburg Hematology Oncology, Lynchburg, Virginia
  - Bon Secours Richmond Community Hospital Medical Oncology Associates at Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours St Francis Medical Center, Midlothian, Virginia
  - Southwest Virginia Regional Cancer Center, Norton, Virginia
  - Bon Secours Richmond Community Hospital Oncology Associates at St. Mary's Hospital, Richmond, Virginia
  - MRCC Auburn, Auburn, Washington
  - MRCC Gig Harbor, Gig Harbor, Washington
  - MRCC Puyallup, Puyallup, Washington
  - MultiCare Health System, Tacoma, Washington
  - MultiCare Institute for Research & Innovation, Tacoma, Washington
  - CAMC Health Education and Research Institute, Charleston, West Virginia
  - West Virginia University, Morgantown, West Virginia
  - Aurora Cancer Care-Southern Lakes, Burlington, Wisconsin
  - Aurora Health Center Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Cancer Care-Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Cancer Care, Milwaukee, Wisconsin
  - Aurora Cancer Care-Milwaukee South, Milwaukee, Wisconsin
  - Aurora St. Lukes Medical Center-Pharmacy Only, Milwaukee, Wisconsin
  - Aurora West Allis Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care, Wauwatosa, Wisconsin
- Canada (5):
  - CIUSSS de l'Est-de-l'Ile-de-Montreal-Hopital-Maisonneuve-Rosemont, Montreal, Quebec
  - Centre Hospitalier d'Universite de Montreal CHUM-Hotel Dieu, Montreal, Quebec
  - SMBD-Jewish General Hospital (MPSG), Montreal, Quebec
  - McGill University Health Centre-Cedars Cancer Centre, Montreal, Quebec
  - CHU de Quebec-Hospital du Saint-Sacrement, Québec, Quebec

REFERENCES:
- [Derived] Perez-Garcia J, Soberino J, Racca F, Gion M, Stradella A, Cortes J. Atezolizumab in the treatment of metastatic triple-negative breast cancer. Expert Opin Biol Ther. 2020 Sep;20(9):981-989. doi: 10.1080/14712598.2020.1769063. Epub 2020 May 25. PMID 32450725